CLINICAL TRIAL: NCT03105336
Title: A Phase 2 Multicenter Study of Axicabtagene Ciloleucel in Subjects With Relapsed/Refractory Indolent Non-Hodgkin Lymphoma (iNHL)
Brief Title: A Study of Axicabtagene Ciloleucel in Participants With Relapsed/Refractory Indolent Non-Hodgkin Lymphoma
Acronym: ZUMA-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-105; 2017-001912-13 (EudraCT Number); 2023-505169-10 (Other: European Medicines Agency)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axicabtagene Ciloleucel (Follicular Lymphoma) (Experimental): Participants with relapsed or refractory (r/r) B-cell indolent non-Hodgkin lymphoma (iNHL) subtype of follicular lymphoma (FL) will receive the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day for 3 days (Day -5 to Day -3).
  * A single infusion at a target dose of 2×10^6 anti-cluster of differentiation 19 (CD19) chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
  Interventions: Biological: Axicabtagene ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Axicabtagene Ciloleucel (Marginal Zone Lymphoma) (Experimental): Participants with r/r B-cell iNHL subtype of marginal zone lymphoma (MZL) will receive the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
  Interventions: Biological: Axicabtagene ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: Axicabtagene ciloleucel — Administered intravenously
  Other Names: Axi-cel; Yescarta®
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously

SUMMARY:
The goal of this study is to assess whether axicabtagene ciloleucel improves the clinical outcome in participants with relapsed or refractory indolent non-Hodgkin lymphoma (r/r) iNHL.

DETAILED DESCRIPTION:
After completing at least 60 months (FL participants) or at least 24 months (MZL participants) of assessments in this study since the initial axicabtagene ciloleucel infusion and after agreement by the Sponsor, participants will transition to a long-term follow-up (LTFU) study, KT-US-982-5968 where they will complete the remainder of the 15 year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Individual has follicular lymphoma (FL) or marginal zone lymphoma (MZL) that has progressed after at least 2 lines of treatment with combination chemoimmunotherapy) (e.g. R-bendamustine, R-CHOP).
* Individual has (measurable disease).
* Individual has no known presence or history of central nervous system (CNS) involvement by lymphoma.
* If individual is on conventional systemic therapy or systemic inhibitory/stimulatory immune checkpoint therapy, individual is able to stop conventional therapy 2 weeks or 5 half-lives, whichever is shorter, or immune checkpoint therapy 3 half-lives prior to planned leukapheresis.
* Individual has Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 and adequate renal, hepatic, pulmonary, and cardiac function
* Individual is not pregnant or breastfeeding (female individuals only) and is willing to use birth control from the time of consent through 12 months following chimeric antigen receptor (CAR) T cell infusion (both male and female individuals).

Key Exclusion Criteria:

* Transformed FL or MZL
* Small lymphocytic lymphoma
* Histological Grade 3b FL
* Individual will have undergone autologous transplant within 6 weeks of planned leukapheresis or has undergone allogeneic transplant.
* Individual has evidence of involvement of the heart by lymphoma or requirement for urgent therapy due to ongoing or impending oncologic emergency (e.g. mass effect, tumor lysis syndrome, etc.)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (19):
- United States (17):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Miami Hospital and Clinics, Miami, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center (URMC), Rochester, New York
  - Ohio State University Medical Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Interim analysis of ZUMA-5: A phase II study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory indolent non-Hodgkin lymphoma (R/R iNHL). Conference Proceedings of the American Society of Clinical Oncology 2020
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Interim analysis of ZUMA-5: A phase II study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory indolent non-Hodgkin lymphoma (R/R iNHL) [Abstract]. Conference Proceedings of the Society of Hematologic Oncology 2020.
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Interim analysis of ZUMA-5: A phase II study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory indolent non-Hodgkin lymphoma (R/R iNHL) [Abstract]. Clinical Lymphoma, Myeloma and Leukemia 2020;20 (1 Suppl):S278.
- [Background] Jacobson C, Chavez JC, Sehgal AR, et al. Primary analysis of Zuma-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL). Blood 2020;136 (1 Suppl):40-41.
- [Background] Chavez JC, Jacobson CA, Sehgal AR, et al. Retreatment with axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory indolent non-Hodgkin lymphoma in ZUMA-5. Blood 2020;136 (1 Suppl):34.
- [Background] Jacobson CA, Chavez JC, Sehgal AR, William BM, Munoz J, Salles G, Munshi PN, Casulo C, Maloney DG, de Vos S, Reshef R, Leslie LA, Yakoub-Agha I, Oluwole OO, Fung HCH, Rosenblatt J, Rossi JM, Goyal L, Plaks V, Yang Y, Vezan R, Avanzi MP, Neelapu SS. Axicabtagene ciloleucel in relapsed or refractory indolent non-Hodgkin lymphoma (ZUMA-5): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2022 Jan;23(1):91-103. doi: 10.1016/S1470-2045(21)00591-X. Epub 2021 Dec 8. PMID 34895487
- [Background] Chavez JC, Jacobson CA, Sehgal A, et al. Updated outcomes with axicabtagene ciloleucel (axi-cel) retreatment (reTx) in patients (pts) with relapsed/refractory (R/R) indolent non-Hodgkin lymphoma (iNHL) in ZUMA-5. J Clin Oncol 2021;39 (15 suppl):7548.
- [Background] Chavez JC, Jacobson CA, Sehgal AR, et al. Retreatment with axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory (r/r) indolent non-hodgkin lymphoma (iNHL) in ZUMA-5 [Oral abstract]. Transplantation and Cellular Therapy 2021;27 (Issue 3, Supplement):S43, ISSN 2666-6367
- [Background] Chavez JC, Jacobson CA, Sehgal AR, et al. Retreatment with axicabtagene ciloleucel in patients with relapsed/refractory indolent non-hodgkin lymphoma in ZUMA-5 [Oral abstract]. British Journal of Heamatology 2021;193. Abstract BSH2021-PO-149.
- [Background] Chavez JC, Jacobson CA, Sehgal AR, et al. Updated outcomes with axicabtagene ciloleucel (axi-cel) retreatment in patients with relapsed/refractory indolent non-Hodgkin lymphoma in ZUMA-5 [Abstract]. European Hematology Association (EHA) 2021:325549.
- [Background] Ghione P, Patel A, Bobillo S, et al. A comparison of clinical outcomes from Zuma-5 (axicabtagene ciloleucel) and the international scholar-5 external control cohort in relapsed/refractory follicular lymphoma (R/R/FL) [Abstract]. European Hematology Association (EHA) Virtual; 2021 09-17 June.
- [Background] Ghione P, Ghesquieres H, Bobillo S, et al. Outcomes in later-lines of therapy for relapsed/refractory follicular lymphoma: results from the international scholar-5 study. Hematological Oncology 2021;39
- [Background] Jacobson CA, Chavez JC, Sehgal A, et al. Outcomes in ZUMA-5 with axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory (R/R) indolent non-Hodgkin lymphoma (iNHL) who had the high-risk feature of progression within 24 months from initiation of first anti-CD20-containing chemoimmunotherapy (POD24). J Clin Oncol 2021a;39 (15 Suppl):7515
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Outcomes in Zuma-5 with axicabtagene ciloleucel in patients with relapsed/refractory indolent non-Hodgkin lymphoma who had the high-risk feature of early progression after first chemoimmunotherapy [Abstract]. European Hematology Association (EHA) Virtual; 2021b 09-17 June.
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Primary analysis of ZUMA-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL) [Oral abstract 69]. Transplantation and Cellular Therapy 2021; 27 (Issue 3, Supplement): S67-S68, ISSN 2666-6367
- [Background] Jacobson CA, Chavez JC, Sehgal AR, et al. Primary analysis of ZUMA-5: A phase 2 study of axicabtagene ciloleucel in patients with relapsed/refractory indolent non-hodgkin lymphoma [Oral abstract]. British Journal of Heamatology 2021, BSH2021-OR-036.
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. Long-term follow-up analysis of ZUMA-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory (R/R) indolent non-Hodgkin lymphoma (iNHL) [Abstract 93]. Blood 2021;138 (1 Suppl)
- [Background] Plaks V, Chou J, Goyal L, et al. Axicabtagene ciloleucel (axi-cel) product attributes and immune biomarkers associated with clinical outcomes in patients (pts) with relapsed/refractory R/R) indolent non-Hodgkin lymphoma (iNHL) in ZUMA-5 [Abstract CT036]. Cancer Res 2021;81 (13 Suppl).
- [Background] Kanters S, Ball G, Kahl B, Wiesinger A, Limbrick-Oldfield EH, Sudhindra A, Snider JT, Patel AR. Clinical outcomes in patients relapsed/refractory after >/=2 prior lines of therapy for follicular lymphoma: a systematic literature review and meta-analysis. BMC Cancer. 2023 Jan 23;23(1):74. doi: 10.1186/s12885-023-10546-6. PMID 36690960
- [Background] Palomba ML, Ghione P, Patel AR, et al. A comparison of clinical outcomes from updated ZUMA-5 (axicabtagene ciloleucel) and the international scholar-5 external control cohort in relapsed/refractory follicular lymphoma (R/R FL) [Abstract PB1571]. Blood 2021;138 (1 Suppl):3543.
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. Long-term follow-up analysis of Zuma-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL) [Abstract 75]. Transplantation and Cellular Therapy 2022;28 (Issue 3, Supplement):S64-S65, ISSN 2666-6367.
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. Long-term analysis of ZUMA-5 phase 2 study of axicabtagene ciloleucel in patients with indolent non-Hodgkin lymphoma [Oral presentation O3-5]. 2022 Japanese Society of Medical Oncology - 19th Scientific Meeting
- [Background] Hatswell AJ, Deighton K, Snider JT, Brookhart MA, Faghmous I, Patel AR. Approaches to Selecting "Time Zero" in External Control Arms with Multiple Potential Entry Points: A Simulation Study of 8 Approaches. Med Decis Making. 2022 Oct;42(7):893-905. doi: 10.1177/0272989X221096070. Epub 2022 May 6. PMID 35514320
- [Background] Ghione P, Palomba ML, Patel AR, Bobillo S, Deighton K, Jacobson CA, Nahas M, Hatswell AJ, Jung AS, Kanters S, Snider JT, Neelapu SS, Ribeiro MT, Brookhart MA, Ghesquieres H, Radford J, Gribben JG. Comparative effectiveness of ZUMA-5 (axi-cel) vs SCHOLAR-5 external control in relapsed/refractory follicular lymphoma. Blood. 2022 Aug 25;140(8):851-860. doi: 10.1182/blood.2021014375. PMID 35679476
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. 3-Year follow-up analysis of ZUMA-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL). Blood 2022;140 (1 Suppl):10380-10383.
- [Background] Oluwole OO, Ray MD, Rosettie KL, Ball G, Jacob J, Bilir SP, Patel AR, Jacobson CA. Cost-Effectiveness of Axicabtagene Ciloleucel for Adult Patients With Relapsed or Refractory Follicular Lymphoma in the United States. Value Health. 2024 Aug;27(8):1030-1038. doi: 10.1016/j.jval.2024.04.003. Epub 2024 Apr 17. PMID 38641058
- [Background] Ghione P, Palomba ML, Ray MD, et al. A 3-year follow-up comparison of clinical outcomes from Zuma-5 (axicabtagene ciloleucel) and the international Scholar-5 external control cohort in relapsed/refractory follicular lymphoma (R/R FL). Blood 2022;140 (1 Suppl):4676-4677.
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. 3-Year follow-up analysis of Zuma-5: A phase 2 study of axicabtagene ciloleucel (axi-cel) in patients (pts) with relapsed/refractory (r/r) indolent non-Hodgkin lymphoma (iNHL) [Abstract 500]. Transplantation and Cellular Therapy 2023;29 (Issue 2, Supplement):S374, ISSN 2666-6367
- [Background] Palomba ML, Ghione P, Patel AR, Nahas M, Beygi S, Hatswell AJ, Kanters S, Limbrick-Oldfield EH, Wade SW, Ray MD, Owen J, Neelapu SS, Gribben J, Radford J, Bobillo S. A 24-month updated analysis of the comparative effectiveness of ZUMA-5 (axi-cel) vs. SCHOLAR-5 external control in relapsed/refractory follicular lymphoma. Expert Rev Anticancer Ther. 2023 Feb;23(2):199-206. doi: 10.1080/14737140.2023.2171994. Epub 2023 Feb 10. PMID 36723678
- [Background] Patel AR, Limbrick-Oldfield EH, Kanters S, et al., The prognostic value of progressing within 24 months of frontline chemoimmunotherapy (POD24) in relapsed/refractory (R/R) follicular lymphoma (FL)-a SCHOLAR-5 analysis. Hematological Oncology 2023;41:376-377.
- [Background] Ray MD, Kanters S, Beygi S, et al. Matching-adjusted indirect comparison of axicabtagene ciloleucel versus mosunetuzumab in relapsed/refractory follicular lymphoma patients after 2 prior systemic treatments. Hematological Oncology 2023;41:522-523
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. Axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory indolent non-Hodgkin lymphoma: 4-year follow-up from the phase 2 ZUMA-5 trial. Blood 2023;142 (1 Suppl):4868.
- [Background] Bachy E, Neelapu SS, Chavez JC, et al. A retrospective intra-patient analysis from ZUMA-5: Axicabtagene ciloleucel (axi-cel) compared with prior standard-of-care therapy in patients with relapsed/refractory follicular lymphoma. Blood 2023;142 (1 Suppl):4865.
- [Background] Gribben JG, Ghione P, Palomba ML, et al. An updated comparison of clinical outcomes from 4-year follow-up of Zuma-5 (axicabtagene ciloleucel) and the international Scholar-5 external control cohort in relapsed/refractory follicular lymphoma. Blood 2023;142 (1 Suppl):4869.
- [Background] Eklund O, Hedlöf Kanje V, Doble B, et al. EE536 Cost-effectiveness of axicabtagene ciloleucel (axi-cel) vs standard of care for adult patients with relapsed or refractory follicular lymphoma as 4TH or later line treatment in Sweden. Value in Health 2023;26 (Issue 12, Supplement):S155, ISSN 1098-3015.
- [Background] Ghione P, Palomba ML, Ray MD, Limbrick-Oldfield EH, Owen J, Kanters S, Bobillo S, Ribiero MT, Jacobson CA, Neelapu SS, Ghesquieres H, Nahas M, Beygi S, Patel AR, Gribben JG. A Comparison of 3-Year Follow-up of ZUMA-5 (Axicabtagene Ciloleucel) With SCHOLAR-5 in Relapsed/Refractory Follicular Lymphoma. Clin Lymphoma Myeloma Leuk. 2024 May;24(5):e191-e195.e6. doi: 10.1016/j.clml.2024.01.011. Epub 2024 Jan 24. PMID 38365528
- [Background] Neelapu SS, Chavez JC, Sehgal AR, Epperla N, Ulrickson M, Bachy E, Munshi PN, Casulo C, Maloney DG, de Vos S, Reshef R, Leslie LA, Oluwole OO, Yakoub-Agha I, Khanal R, Rosenblatt J, Korn R, Peng W, Lui C, Wulff J, Shen R, Poddar S, Jung AS, Miao H, Beygi S, Jacobson CA. Three-year follow-up analysis of axicabtagene ciloleucel in relapsed/refractory indolent non-Hodgkin lymphoma (ZUMA-5). Blood. 2024 Feb 8;143(6):496-506. doi: 10.1182/blood.2023021243. PMID 37879047
- [Background] Oluwole OO, Ray MD, Zur RM, Ferrufino CP, Doble B, Patel AR, Bilir SP. Cost-effectiveness of treating relapsed or refractory 3L+ follicular lymphoma with axicabtagene ciloleucel vs mosunetuzumab in the United States. Front Immunol. 2024 May 24;15:1393939. doi: 10.3389/fimmu.2024.1393939. eCollection 2024. PMID 38855109
- [Background] Ray MD, Kanters S, Beygi S, Best T, Wulff J, Limbrick-Oldfield E, Patel AR, Oluwole OO. Matching-Adjusted Indirect Comparisons of Axicabtagene Ciloleucel to Mosunetuzumab for the Treatment of Relapsed/Refractory Follicular Lymphoma. Transplant Cell Ther. 2024 Sep;30(9):885.e1-885.e11. doi: 10.1016/j.jtct.2024.06.016. Epub 2024 Jun 19. PMID 38901633
- [Background] Neelapu SS, Chavez JC, Sehgal AR, et al. 5-year follow-up analysis from ZUMA-5: A phase 2 trial of axicabtagene ciloleucel (axi-cel) in patients with relapsed/refractory indolent non-Hodgkin lymphoma. Blood 2024;144 (1 Suppl):864.
- [Background] Poddar S, Yan J, Tiwari G, et al. Impact of inflammation, tumor and product attributes on clinical outcomes in patients with relapsed/refractory follicular lymphoma treated with axicabtagene ciloleucel. Blood 2024;144 (1 Suppl):4368
- [Background] Limbrick-Oldfield EH, Kanters S, Ray MD, Best T, Palivela M, Beygi S, Patel AR, Gribben JG, Ghione P. The prognostic value of POD24 in relapsed/refractory follicular lymphoma-A SCHOLAR-5 analysis. EJHaem. 2025 Feb 6;6(1):e1104. doi: 10.1002/jha2.1104. eCollection 2025 Feb. PMID 39917356
- [Derived] Neelapu SS, Chavez JC, Sehgal AR, Epperla N, Ulrickson ML, Bachy E, Munshi PN, Casulo C, Maloney DG, de Vos S, Reshef R, Leslie LA, Oluwole OO, Yakoub-Agha I, Khanal R, Rosenblatt JD, Wulff J, Shen RR, Zhang W, Poddar S, Miao H, Nikolajeva O, Jacobson CA. Five-Year Follow-Up Analysis of ZUMA-5: Axicabtagene Ciloleucel in Relapsed/Refractory Indolent Non-Hodgkin Lymphoma. J Clin Oncol. 2025 Nov 20;43(33):3573-3577. doi: 10.1200/JCO-25-00668. Epub 2025 Oct 16. PMID 41100801
- [Derived] Poddar S, Yan J, Tiwari G, Rinchai D, Budka J, Zhang W, Peng W, Salunkhe S, Davis M, Song Q, Beygi S, Miao H, Mattie M, Shen RS, Jacobson CA, Bedognetti D, Filosto S, Neelapu SS. Clinical, tumor, and product features associated with outcomes after axicabtagene ciloleucel therapy in follicular lymphoma. J Clin Invest. 2025 Aug 15;135(16):e181893. doi: 10.1172/JCI181893. eCollection 2025 Aug 15. PMID 40536814
- [Derived] Chartier M, Filosto S, Peyret T, Chiney M, Milletti F, Budka J, Ndi A, Dong J, Vardhanabhuti S, Mao D, Duffull S, Dodds M, Shen R. Investigating the Influence of Covariates on Axicabtagene Ciloleucel (axi-cel) Kinetics in Patients with Non-Hodgkin's Lymphoma. Clin Pharmacokinet. 2024 Sep;63(9):1283-1299. doi: 10.1007/s40262-024-01413-z. Epub 2024 Sep 6. PMID 39240498
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and France.
Pre-assignment Details: 189 participants were screened. A total of 159 participants were enrolled. However, one participant discontinued the study as the participant did not meet study condition eligibility criteria (was diagnosed with diffuse large B-cell lymphoma (DLBCL)). So, 158 participants were considered in the Full Analysis Set (FAS = all enrolled participants).
Groups:
- Axicabtagene Ciloleucel (Follicular Lymphoma): Participants with relapsed or refractory (r/r) B-cell indolent non-Hodgkin lymphoma (iNHL) subtype of follicular lymphoma (FL) received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day intravenously (IV) and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-cluster of differentiation 19 (CD19) chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
- Axicabtagene Ciloleucel (Marginal Zone Lymphoma): Participants with r/r B-cell iNHL subtype of marginal zone lymphoma (MZL) received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day IV and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
Period: Overall Study
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Started | 127 | 31
Completed | 0 | 0
Not Completed | 127 | 31
Not completed — Rollover to Longterm Follow-up Study Criteria | 61 | 15
Not completed — Death | 40 | 8
Not completed — Lost to Follow-up | 13 | 2
Not completed — Subject Withdrawal of Consent from Further Follow-up | 7 | 3
Not completed — Reason Not Specified | 3 | 3
Not completed — Investigator Decision | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was defined as all participants treated with any dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma) | Total
Number analyzed (Participants) | 124 | 28 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 15 | 101
  >=65 years | 38 | 13 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.9) | 63 (9.6) | 60.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 15 | 66
  Male | 73 | 13 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 118 | 24 | 142
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 115 | 25 | 140
  Race: Black or African American | 4 | 2 | 6
  Race: Other or More Than One Race | 3 | 1 | 4
  Race: Asian | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 114 | 28 | 142
  France | 10 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response Per the Lugano Classification by Central Assessment
Description: OR:CR (complete metabolic response (CMR)+complete radiological response (CRR))+PR (partial MR response (PMR) +partial RR(PRR)).CMR: score 1(no uptake above background)/2(uptake≤mediastinum)/3(uptake >mediastinum but ≤liver)with/without a residual mass on positron emission tomography 5-point scale;no new lesions,CRR:target nodes/nodal masses regressed to ≤1.5 cm in longest transverse diameter of lesion (LDi);no extralymphatic sites of disease;absent non-measured lesion(NMLs);organ enlargement regress to normal; no new sites;bone marrow normal by morphology.PMR:score 4(uptake moderately>liver)/5(uptake markedly>liver, new lesions) with reduced uptake compared with baseline and residual mass;no new lesions;responding disease at interim/residual disease at end of treatment.PRR:≥50% decrease in sum of product of diameters up to 6 target nodes and extra-nodal sites;absent/normal,regressed,but no increase of NMLs;spleen regressed by>50% in length beyond normal. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set with available data were analyzed. Full Analysis Set consisted of all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Axicabtagene Ciloleucel (Follicular Lymphoma): Participants with r/r B-cell iNHL subtype of FL received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day IV and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
- Axicabtagene Ciloleucel (Marginal Zone Lymphoma): Participants with r/r B-cell iNHL subtype of MZL received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day IV and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 29
percentage of participants | 92 [86 to 96] | 69 [49 to 85]

2. Secondary Outcome: Percentage of Participants With CR Per the Lugano Classification by Central Assessment
Description: CR is defined in outcome measure (OM)#1. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 29
percentage of participants | 78 [70 to 85] | 52 [33 to 71]

3. Secondary Outcome: ORR: Percentage of Participants With OR Per the Lugano Classification by Central Assessment Among Participants With 3 or More Lines of Prior Therapy
Description: OR was defined as percentage of participants with CR + PR per the Lugano Classification for participants with 3 or more lines of prior therapy. CR and PR are defined in OM#1. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants with 3 or more lines of prior therapy in the Full Analysis Set with available data were analyzed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 80 | 20
percentage of participants | 91 [83 to 96] | 75 [51 to 91]

4. Secondary Outcome: Percentage of Participants With CR Per Lugano Classification by Central Assessment Among Participants With 3 or More Lines of Prior Therapy
Description: CR is defined as OM#1. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants with 3 or more lines of prior therapy in the Full Analysis Set with available data were analyzed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 80 | 20
percentage of participants | 79 [68 to 87] | 60 [36 to 81]

5. Secondary Outcome: ORR: Percentage of Participants With OR Per the Lugano Classification by Investigator Assessment
Description: OR was defined as percentage of participants with CR + PR per the Lugano Classification. CR and PR are defined in OM#1. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 31
percentage of participants | 94 [88 to 97] | 77 [59 to 90]

6. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) Per the Lugano Classification by Central Assessment
Description: BOR was defined as percentage of participants with CR, PR, stable disease(SD), disease progression(PD), non-evaluable(NE), undefined/no disease or not done as best response to treatment by the Lugano Classification. CR and PR defined in OM#1. SD/no metabolic response(NMR):score 4(uptake moderately greater than (>) liver) or 5(uptake markedly>liver and/ or new lesions) with no significant change in fluorodeoxyglucose(FDG) uptake compared to baseline(screening), at interim time point or end of treatment; no new sites of disease should be observed. PD:score 4(uptake moderately>liver) or 5(uptake markedly>liver and/or new lesions) with an increase in intensity of uptake from baseline; new FDG-avid foci consistent with lymphoma at interim or end of treatment assessment; new FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation); new or recurrent FDG-avid foci in bone marrow. Not done:no assessment at time of analysis. Percentages were rounded off.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set with available data were analyzed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 29
percentage of participants
  CR | 78 [70 to 85] | 52 [33 to 71]
  PR | 14 [9 to 21] | 17 [6 to 36]
  SD | 4 [1 to 9] | 0 [0 to 12]
  PD | 0 [0 to 3] | 3 [0 to 18]
  Non-evaluable | 0 [0 to 3] | 0 [0 to 12]
  Undefined/ No Disease | 1 [0 to 4] | 10 [2 to 27]
  Not Done | 3 [1 to 8] | 17 [6 to 36]

7. Secondary Outcome: Percentage of Participants With BOR Per the Lugano Classification by Investigator Assessment
Description: BOR was defined as the percentage of participants with CR, PR, stable disease (SD), PD, NE (not evaluable) or not done as best response to treatment by the Lugano Classification. CR and PR are defined in OM#1. SD, PD and not done are defined in OM#6. Percentages were rounded off.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 31
percentage of participants
  CR | 79 [71 to 85] | 65 [45 to 81]
  PR | 15 [9 to 22] | 13 [4 to 30]
  SD | 2 [0 to 6] | 10 [2 to 26]
  PD | 2 [0 to 6] | 3 [0 to 17]
  NE | 0 [0 to 3] | 0 [0 to 11]
  Not Done | 3 [1 to 8] | 10 [2 to 26]

8. Secondary Outcome: Duration of Response (DOR) by Central Assessment
Description: DOR was defined only for participants who experienced an OR (CR and PR) and was the time from the first objective response to disease progression or disease-related death, whichever came first. CR and PR are defined in OM#1. PD is defined in OM#6.
  Kaplan-Meier (KM) estimates were used for analysis.
Time Frame: Up to 85.6 months
Population: Participants with OR in the Full Analysis Set with available data were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 117 | 20
months | 38.6 [NA to NA] — Lower and upper limit of confidence intervals (CI) could not be estimated due to limited number of events and censoring. The Median was estimated because the longest observed participant event crossed 50%. | NA [8.2 to NA] — Data for median and upper limit of CI were not estimable due to low number of participants with events.

9. Secondary Outcome: DOR by Investigator Assessment
Description: DOR was defined only for participants who experienced an OR (CR and PR) and was the time from the first objective response to disease progression or disease-related death, whichever came first. Definitions for CR, PR are defined in OM#1. PD is defined in OM#6.
  KM estimates were used for analysis.
Time Frame: Up to 85.6 months
Population: Participants with OR in Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 119 | 24
months | 60.4 [36.6 to NA] — Data for upper limit of CI was not estimable due to low number of participants with events. | NA [13.9 to NA] — Data for median and upper limit of CI was not estimable due to low number of participants with events.

10. Secondary Outcome: Progression-free Survival (PFS) Per Lugano Classification by Central Assessment
Description: PFS was defined as the time from the axicabtagene ciloleucel infusion date to the date of disease progression per Lugano classification or death from any cause. PD is defined in OM 6. KM estimates were used for analysis.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 29
months | 40.2 [28.9 to NA] — Data for upper limit of CI was not estimable due to low number of participants with events. | 18.3 [12.1 to NA] — Data for median and upper limit of CI was not estimable due to low number of participants with events.

11. Secondary Outcome: PFS Per Lugano Classification by Investigator Assessment
Description: as for outcome 10
Time Frame: Up to 85.6 months
Population: Participants in Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 31
months | 58.2 [30.9 to NA] — Data for upper limit of CI was not estimable due to low number of participants with events. | NA [12.4 to NA] — Data for median and upper limit of CI was not estimable due to low number of participants with events.

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from axicabtagene ciloleucel infusion to the date of death. KM estimates were used for analysis.
Time Frame: Up to 85.6
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 31
months | NA [NA to NA] — Data for median, lower, and upper limits of CI were not estimable due to low number of participants with events | NA [NA to NA] — Data for median, lower, and upper limits of CI were not estimable due to low number of participants with events

13. Secondary Outcome: Time to Next Therapy
Description: Time from axicabtagene ciloleucel infusion date to the start of the subsequent new lymphoma therapy or death from any cause. KM estimates were used for analysis.
Time Frame: Up to 85.6 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 127 | 31
months | NA [37.8 to NA] — Data for median and upper limit of CI were not estimable due to low number of participants with events. | NA [12.1 to NA] — Data for median and upper limit of CI were not estimable due to low number of participants with events.

14. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: TEAE was defined as any adverse event with onset on or after the start of treatment. Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
percentage of participants | 99 | 100

15. Secondary Outcome: Percentage of Participants With Increase in Laboratory Values Reported as Grade 3 or Higher
Description: Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
percentage of participants
  Grade 3 or Higher Increase in Hemoglobin (mmol/L) | 0 | 0
  Grade 3 or Higher Increase in Leukocytes (10^9/L) | 1 | 0
  Grade 3 or Higher Increase in Lymphocytes (10^9/L) | 0 | 0
  Grade 3 or Higher Increase in Alanine Aminotransferase (U/L) | 6 | 21
  Grade 3 or Higher Increase in Alkaline Phosphatase (U/L) | 0 | 4
  Grade 3 or Higher Increase in Aspartate Aminotransferase (U/L) | 4 | 11
  Grade 3 or Higher Increase in Bilirubin (umol/L) | 4 | 11
  Grade 3 or Higher Increase in Calcium (mmol/L) | 1 | 0
  Grade 3 or Higher Increase in Creatinine (umol/L) | 1 | 0
  Grade 3 or Higher Increase in Direct Bilirubin (umol/L) | 2 | 11
  Grade 3 or Higher Increase in Glucose (mmol/L) | 9 | 21
  Grade 3 or Higher Increase in Magnesium (mmol/L) | 3 | 4
  Grade 3 or Higher Increase in Potassium (mmol/L) | 1 | 0
  Grade 3 or Higher Increase in Sodium (mmol/L) | 0 | 0
  Grade 3 or Higher Increase in Urate (mmol/L) | 13 | 25

16. Secondary Outcome: Percentage of Participants With Decrease in Laboratory Values Reported as Grade 3 or Higher
Description: Percentages were rounded-off.
Time Frame: Up to 85.6 months
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
percentage of participants
  Grade 3 or Higher Decrease in Hemoglobin (mmol/L) | 33 | 39
  Grade 3 or Higher Decrease in Leukocytes (10^9/L) | 94 | 93
  Grade 3 or Higher Decrease in Lymphocytes (10^9/L) | 99 | 100
  Grade 3 or Higher Decrease in Neutrophils (10^9/L) | 92 | 96
  Grade 3 or Higher Decrease in Platelets (10^9/L) | 35 | 32
  Grade 3 or Higher Decrease in Albumin (g/L) | 2 | 4
  Grade 3 or Higher Decrease in Calcium (mmol/L) | 10 | 7
  Grade 3 or Higher Decrease in Glucose (mmol/L) | 0 | 0
  Grade 3 or Higher Decrease in Magnesium (mmol/L) | 0 | 0
  Grade 3 or Higher Decrease in Phosphate (mmol/L) | 23 | 39
  Grade 3 or Higher Decrease in Potassium (mmol/L) | 4 | 7
  Grade 3 or Higher Decrease in Sodium (mmol/L) | 9 | 18

17. Secondary Outcome: Percentage of Participants With Antibodies Against Anti-CD19 Chimeric Antigen Receptor (CAR) T Cells
Time Frame: Up to 85.6 months
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
percentage of participants | 0 | 0

18. Secondary Outcome: Levels of Anti-CD19 CAR T Cells in Blood
Time Frame: Day 7, Week 2, Week 4, Month 3, Month 6, Month 12, Month 18 and Month 24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
cells/μL
  Day 7 | 101.49 (220.01) | 120.07 (394.91)
  Week 2: number analyzed (Participants) | 112 | 26
  Week 2 | 41.45 (63.65) | 90.76 (128.63)
  Week 4: number analyzed (Participants) | 117 | 27
  Week 4 | 7.52 (19.85) | 14.03 (23.43)
  Month 3: number analyzed (Participants) | 114 | 24
  Month 3 | 0.78 (1.91) | 0.52 (0.51)
  Month 6: number analyzed (Participants) | 106 | 24
  Month 6 | 3.49 (28.89) | 0.68 (1.90)
  Month 12: number analyzed (Participants) | 86 | 15
  Month 12 | 1.00 (5.65) | 0.23 (0.43)
  Month 18: number analyzed (Participants) | 66 | 17
  Month 18 | 0.47 (1.51) | 0.42 (0.77)
  Month 24: number analyzed (Participants) | 65 | 16
  Month 24 | 0.36 (0.84) | 0.88 (2.09)

19. Secondary Outcome: Levels of Serum C-Reactive Protein (CRP)
Time Frame: Baseline (at enrollment), predose: Day 0, postdose: Day 3, Day 7, Week 2, Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 123 | 28
mg/L
  Serum CRP on Baseline: number analyzed (Participants) | 122 | 28
  Serum CRP on Baseline | 22.36 (40.60) | 19.87 (28.62)
  Serum CRP on Day 0: number analyzed (Participants) | 121 | 28
  Serum CRP on Day 0 | 29.30 (47.35) | 32.94 (42.50)
  Serum CRP on Day 3: number analyzed (Participants) | 106 | 27
  Serum CRP on Day 3 | 72.50 (91.76) | 66.73 (92.82)
  Serum CRP on Day 7 | 59.45 (79.24) | 77.79 (91.86)
  Serum CRP on Week 2: number analyzed (Participants) | 113 | 26
  Serum CRP on Week 2 | 9.07 (19.70) | 13.59 (42.20)
  Serum CRP on Week 4: number analyzed (Participants) | 118 | 28
  Serum CRP on Week 4 | 7.84 (33.76) | 9.86 (43.46)

20. Secondary Outcome: Levels of Serum Ferritin, Serum ICAM-1, Serum IL-2 R Alpha, Serum Perforin and Serum VCAM-1
Description: Serum analytes: Serum Ferritin, Serum intercellular adhesion molecule-1 (ICAM-1), Serum interleukin-2 receptor (IL-2 R) alpha, Serum Perforin and Serum vascular cell adhesion molecule-1 (VCAM-1).
Time Frame: Baseline (at enrollment), predose: Day 0, postdose: Day 3, Day 7, Week 2, Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
ng/L
  Serum Ferritin on Baseline: number analyzed (Participants) | 122 | 28
  Serum Ferritin on Baseline | 330.54 (398.03) | 207.63 (218.42)
  Serum Ferritin on Day 0: number analyzed (Participants) | 121 | 28
  Serum Ferritin on Day 0 | 503.99 (502.07) | 398.49 (337.82)
  Serum Ferritin on Day 3: number analyzed (Participants) | 106 | 27
  Serum Ferritin on Day 3 | 541.51 (457.18) | 487.39 (414.90)
  Serum Ferritin on Day 7: number analyzed (Participants) | 123 | 28
  Serum Ferritin on Day 7 | 779.75 (782.98) | 1820.38 (4837.56)
  Serum Ferritin on Week 2: number analyzed (Participants) | 113 | 26
  Serum Ferritin on Week 2 | 741.76 (787.70) | 959.49 (1546.07)
  Serum Ferritin on Week 4: number analyzed (Participants) | 118 | 28
  Serum Ferritin on Week 4 | 528.83 (605.94) | 478.47 (459.54)
  Serum ICAM-1 on Baseline: number analyzed (Participants) | 122 | 28
  Serum ICAM-1 on Baseline | 876.99 (833.80) | 709.71 (430.14)
  Serum ICAM-1 on Day 0: number analyzed (Participants) | 121 | 28
  Serum ICAM-1 on Day 0 | 834.87 (854.35) | 642.60 (365.92)
  Serum ICAM-1 on Day 3: number analyzed (Participants) | 106 | 27
  Serum ICAM-1 on Day 3 | 964.45 (904.79) | 792.47 (621.84)
  Serum ICAM-1 on Day 7: number analyzed (Participants) | 123 | 28
  Serum ICAM-1 on Day 7 | 924.99 (846.56) | 934.02 (618.96)
  Serum ICAM-1 on Week 2: number analyzed (Participants) | 113 | 26
  Serum ICAM-1 on Week 2 | 695.15 (605.03) | 696.77 (438.71)
  Serum ICAM-1 on Week 4: number analyzed (Participants) | 118 | 28
  Serum ICAM-1 on Week 4 | 671.32 (656.46) | 614.92 (487.67)
  Serum IL-2 R alpha on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-2 R alpha on Baseline | 8.52 (12.15) | 5.62 (7.50)
  Serum IL-2 R alpha on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-2 R alpha on Day 0 | 8.39 (9.10) | 4.91 (4.12)
  Serum IL-2 R alpha on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-2 R alpha on Day 3 | 9.96 (11.53) | 7.31 (5.68)
  Serum IL-2 R alpha on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-2 R alpha on Day 7 | 14.42 (15.10) | 19.78 (20.82)
  Serum IL-2 R alpha on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-2 R alpha on Week 2 | 7.16 (8.27) | 10.40 (12.26)
  Serum IL-2 R alpha on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-2 R alpha on Week 4 | 3.39 (3.34) | 4.02 (3.67)
  Serum Perforin on Baseline: number analyzed (Participants) | 122 | 28
  Serum Perforin on Baseline | 13.26 (7.20) | 13.58 (18.33)
  Serum Perforin on Day 0: number analyzed (Participants) | 121 | 28
  Serum Perforin on Day 0 | 2.56 (1.85) | 3.30 (9.11)
  Serum Perforin on Day 3: number analyzed (Participants) | 106 | 27
  Serum Perforin on Day 3 | 3.87 (3.36) | 4.71 (13.53)
  Serum Perforin on Day 7 | 8.49 (10.54) | 6.60 (7.99)
  Serum Perforin on Week 2: number analyzed (Participants) | 113 | 26
  Serum Perforin on Week 2 | 8.06 (6.90) | 6.01 (6.77)
  Serum Perforin on Week 4: number analyzed (Participants) | 118 | 28
  Serum Perforin on Week 4 | 14.56 (11.92) | 12.32 (12.08)
  Serum VCAM-1 on Baseline: number analyzed (Participants) | 122 | 28
  Serum VCAM-1 on Baseline | 1499.37 (1637.98) | 1282.81 (1232.76)
  Serum VCAM-1 on Day 0: number analyzed (Participants) | 121 | 28
  Serum VCAM-1 on Day 0 | 1182.41 (1166.58) | 931.58 (709.94)
  Serum VCAM-1 on Day 3: number analyzed (Participants) | 106 | 27
  Serum VCAM-1 on Day 3 | 1213.84 (962.38) | 1044.96 (870.11)
  Serum VCAM-1 on Day 7: number analyzed (Participants) | 123 | 28
  Serum VCAM-1 on Day 7 | 1224.58 (1069.13) | 1209.51 (780.31)
  Serum VCAM-1 on Week 2: number analyzed (Participants) | 113 | 26
  Serum VCAM-1 on Week 2 | 891.64 (726.10) | 977.88 (919.47)
  Serum VCAM-1 on Week 4: number analyzed (Participants) | 118 | 28
  Serum VCAM-1 on Week 4 | 981.67 (879.87) | 930.89 (885.51)

21. Secondary Outcome: Levels of Serum CXCL10, Serum Granzyme B, Serum IFN-gamma, Serum IL-1 RA, Serum IL-2, Serum IL-6, Serum IL-7, Serum IL-8, Serum IL-10, Serum IL-15, Serum TNF Alpha
Description: Serum analytes: Serum CXCL10, Serum Granzyme B, Serum interferon (IFN)-gamma, Serum IL-1 receptor antagonist (RA), Serum IL-2, Serum IL-6, Serum IL-7, Serum IL-8, Serum IL-10, Serum IL-15, Serum tumor necrosis factor (TNF) Alpha.
Time Frame: Baseline (at enrollment), predose: Day 0, postdose: Day 3, Day 7, Week 2, Week 4
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Axicabtagene Ciloleucel (Follicular Lymphoma) | Axicabtagene Ciloleucel (Marginal Zone Lymphoma)
Number analyzed (Participants) | 124 | 28
pg/mL
  Serum CXCL10 on Baseline: number analyzed (Participants) | 122 | 28
  Serum CXCL10 on Baseline | 466.32 (339.00) | 634.56 (539.17)
  Serum CXCL10 on Day 0: number analyzed (Participants) | 121 | 28
  Serum CXCL10 on Day 0 | 499.16 (334.85) | 763.99 (569.42)
  Serum CXCL10 on Day 3: number analyzed (Participants) | 106 | 27
  Serum CXCL10 on Day 3 | 712.31 (543.76) | 962.96 (611.23)
  Serum CXCL10 on Day 7: number analyzed (Participants) | 123 | 28
  Serum CXCL10 on Day 7 | 841.62 (572.80) | 1630.98 (563.40)
  Serum CXCL10 on Week 2: number analyzed (Participants) | 113 | 26
  Serum CXCL10 on Week 2 | 474.45 (371.95) | 798.28 (631.80)
  Serum CXCL10 on Week 4: number analyzed (Participants) | 118 | 28
  Serum CXCL10 on Week 4 | 623.87 (535.45) | 964.92 (640.57)
  Serum Granzyme B on Baseline: number analyzed (Participants) | 122 | 28
  Serum Granzyme B on Baseline | 3.58 (9.68) | 121.49 (623.76)
  Serum Granzyme B on Day 0: number analyzed (Participants) | 121 | 28
  Serum Granzyme B on Day 0 | 2.95 (7.86) | 46.36 (234.23)
  Serum Granzyme B on Day 3: number analyzed (Participants) | 106 | 27
  Serum Granzyme B on Day 3 | 6.53 (11.03) | 74.28 (348.53)
  Serum Granzyme B on Day 7 | 76.29 (494.66) | 52.87 (68.63)
  Serum Granzyme B on Week 2: number analyzed (Participants) | 113 | 26
  Serum Granzyme B on Week 2 | 2.73 (5.67) | 27.21 (102.65)
  Serum Granzyme B on Week 4: number analyzed (Participants) | 118 | 28
  Serum Granzyme B on Week 4 | 3.14 (5.15) | 17.00 (39.90)
  Serum IFN-gamma on Baseline: number analyzed (Participants) | 122 | 28
  Serum IFN-gamma on Baseline | 9.25 (7.17) | 30.29 (83.67)
  Serum IFN-gamma on Day 0: number analyzed (Participants) | 121 | 28
  Serum IFN-gamma on Day 0 | 11.20 (16.17) | 54.04 (140.40)
  Serum IFN-gamma on Day 3: number analyzed (Participants) | 106 | 27
  Serum IFN-gamma on Day 3 | 157.13 (326.44) | 292.67 (531.54)
  Serum IFN-gamma on Day 7: number analyzed (Participants) | 123 | 28
  Serum IFN-gamma on Day 7 | 139.82 (359.84) | 674.34 (792.31)
  Serum IFN-gamma on Week 2: number analyzed (Participants) | 113 | 26
  Serum IFN-gamma on Week 2 | 25.98 (48.82) | 27.16 (37.43)
  Serum IFN-gamma on Week 4: number analyzed (Participants) | 118 | 28
  Serum IFN-gamma on Week 4 | 23.96 (37.04) | 56.72 (108.10)
  Serum IL-1 RA on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-1 RA on Baseline | 584.66 (400.47) | 627.95 (467.39)
  Serum IL-1 RA on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-1 RA on Day 0 | 677.50 (743.22) | 960.41 (1342.30)
  Serum IL-1 RA on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-1 RA on Day 3 | 703.79 (772.95) | 848.20 (757.98)
  Serum IL-1 RA on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-1 RA on Day 7 | 1125.80 (1316.88) | 2492.85 (2895.93)
  Serum IL-1 RA on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-1 RA on Week 2 | 591.72 (764.19) | 854.68 (1693.69)
  Serum IL-1 RA on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-1 RA on Week 4 | 653.88 (1197.23) | 1106.94 (1935.55)
  Serum IL-2 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-2 on Baseline | 1.03 (0.53) | 1.12 (0.90)
  Serum IL-2 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-2 on Day 0 | 1.20 (1.22) | 1.16 (1.09)
  Serum IL-2 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-2 on Day 3 | 8.01 (13.08) | 12.43 (34.49)
  Serum IL-2 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-2 on Day 7 | 1.67 (2.55) | 2.99 (3.78)
  Serum IL-2 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-2 on Week 2 | 0.95 (0.48) | 0.93 (0.18)
  Serum IL-2 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-2 on Week 4 | 0.95 (0.50) | 1.10 (1.06)
  Serum IL-6 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-6 on Baseline | 2.71 (2.90) | 5.08 (8.11)
  Serum IL-6 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-6 on Day 0 | 2.42 (2.27) | 4.14 (5.39)
  Serum IL-6 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-6 on Day 3 | 59.30 (185.89) | 103.93 (281.61)
  Serum IL-6 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-6 on Day 7 | 67.49 (197.95) | 206.75 (282.31)
  Serum IL-6 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-6 on Week 2 | 20.01 (92.15) | 33.00 (66.24)
  Serum IL-6 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-6 on Week 4 | 31.02 (122.14) | 58.84 (169.85)
  Serum IL-7 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-7 on Baseline | 15.99 (7.89) | 15.30 (7.13)
  Serum IL-7 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-7 on Day 0 | 27.65 (9.62) | 28.31 (10.15)
  Serum IL-7 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-7 on Day 3 | 26.50 (10.22) | 27.24 (10.82)
  Serum IL-7 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-7 on Day 7 | 23.42 (11.28) | 23.28 (11.69)
  Serum IL-7 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-7 on Week 2 | 27.25 (14.13) | 26.38 (16.52)
  Serum IL-7 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-7 on Week 4 | 18.45 (8.92) | 20.30 (10.52)
  Serum IL-8 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-8 on Baseline | 13.59 (15.09) | 13.71 (9.11)
  Serum IL-8 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-8 on Day 0 | 21.12 (33.53) | 42.71 (129.39)
  Serum IL-8 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-8 on Day 3 | 60.27 (126.84) | 80.86 (154.41)
  Serum IL-8 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-8 on Day 7 | 45.79 (86.38) | 37.47 (30.74)
  Serum IL-8 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-8 on Week 2 | 16.08 (17.14) | 41.41 (117.98)
  Serum IL-8 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-8 on Week 4 | 20.36 (68.72) | 18.90 (13.80)
  Serum IL-10 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-10 on Baseline | 2.85 (3.76) | 5.11 (6.72)
  Serum IL-10 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-10 on Day 0 | 1.93 (2.29) | 1.89 (2.18)
  Serum IL-10 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-10 on Day 3 | 9.34 (17.60) | 7.39 (10.14)
  Serum IL-10 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-10 on Day 7 | 15.01 (34.55) | 20.32 (20.70)
  Serum IL-10 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-10 on Week 2 | 2.06 (4.64) | 3.42 (4.88)
  Serum IL-10 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-10 on Week 4 | 1.10 (1.31) | 1.65 (2.08)
  Serum IL-15 on Baseline: number analyzed (Participants) | 122 | 28
  Serum IL-15 on Baseline | 2.70 (2.69) | 2.59 (1.42)
  Serum IL-15 on Day 0: number analyzed (Participants) | 121 | 28
  Serum IL-15 on Day 0 | 31.06 (13.55) | 33.89 (16.32)
  Serum IL-15 on Day 3: number analyzed (Participants) | 106 | 27
  Serum IL-15 on Day 3 | 35.27 (19.66) | 43.43 (37.40)
  Serum IL-15 on Day 7: number analyzed (Participants) | 123 | 28
  Serum IL-15 on Day 7 | 18.73 (9.77) | 25.22 (15.38)
  Serum IL-15 on Week 2: number analyzed (Participants) | 113 | 26
  Serum IL-15 on Week 2 | 10.30 (5.90) | 12.92 (8.28)
  Serum IL-15 on Week 4: number analyzed (Participants) | 118 | 28
  Serum IL-15 on Week 4 | 4.98 (3.52) | 7.41 (5.21)
  Serum TNF Alpha on Baseline: number analyzed (Participants) | 122 | 28
  Serum TNF Alpha on Baseline | 7.26 (7.87) | 6.73 (7.86)
  Serum TNF Alpha on Day 0: number analyzed (Participants) | 121 | 28
  Serum TNF Alpha on Day 0 | 3.32 (2.62) | 3.08 (1.68)
  Serum TNF Alpha on Day 3: number analyzed (Participants) | 106 | 27
  Serum TNF Alpha on Day 3 | 3.95 (2.68) | 4.90 (4.59)
  Serum TNF Alpha on Day 7: number analyzed (Participants) | 123 | 28
  Serum TNF Alpha on Day 7 | 3.93 (3.10) | 5.97 (4.09)
  Serum TNF Alpha on Week 2: number analyzed (Participants) | 113 | 26
  Serum TNF Alpha on Week 2 | 2.84 (6.01) | 2.74 (2.30)
  Serum TNF Alpha on Week 4: number analyzed (Participants) | 118 | 28
  Serum TNF Alpha on Week 4 | 2.36 (1.65) | 3.03 (2.13)

ADVERSE EVENTS:
Time Frame: Up to 85.6 months
Description: All-cause mortality included Full Analysis Set, that included all enrolled participants.
  Adverse events Safety Analysis Set, that included all participants treated with any dose of study drug.
  Retreatment arms included the Safety-Retreatment Analysis Set, that included all participants with re-treatment of Axicabtagene Ciloleucel from Safety Analysis Set.
Groups:
- Axicabtagene Ciloleucel: Follicular Lymphoma: Participants with r/r B-cell iNHL subtype of FL received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day IV and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
- Axicabtagene Ciloleucel: Marginal Zone Lymphoma: Participants with r/r B-cell iNHL subtype of MZL received the following treatment during the study:
  * A conditioning chemotherapy regimen of fludarabine 30 mg/m^2/day IV and cyclophosphamide 500 mg/m^2/day IV for 3 days (Day -5 to Day -3).
  * A single IV infusion at a target dose of 2×10^6 anti-CD19 CAR transduced autologous T cells/kg on Day 0.
- Axicabtagene Ciloleucel: Retreatment (FL): Participants with r/r iNHL subtype of FL who achieved a response of PR or better at the 3-month disease assessment, but subsequently experienced disease progression, received a second course of conditioning chemotherapy and IV infusion of 2 × 10^6 anti-CD19 CAR transduced autologous T, once at any time during the study.
- Axicabtagene Ciloleucel: Retreatment (MZL): Participants with r/r iNHL subtype of MZL who achieved a response of PR or better at the 3-month disease assessment, but subsequently experienced disease progression, received a second course of conditioning chemotherapy and IV infusion of 2 × 10^6 anti-CD19 CAR transduced autologous T, once at any time during the study.
Arm/Group | Axicabtagene Ciloleucel: Follicular Lymphoma | Axicabtagene Ciloleucel: Marginal Zone Lymphoma | Axicabtagene Ciloleucel: Retreatment (FL) | Axicabtagene Ciloleucel: Retreatment (MZL)
All-Cause Mortality (participants affected / at risk) | 36/127 | 8/31 | 5/14 | 0/2
Serious Adverse Events (participants affected / at risk) | 65/124 | 19/28 | 5/14 | 1/2
Other Adverse Events (participants affected / at risk) | 123/124 | 28/28 | 13/14 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel: Follicular Lymphoma (N=124) | Axicabtagene Ciloleucel: Marginal Zone Lymphoma (N=28) | Axicabtagene Ciloleucel: Retreatment (FL) (N=14) | Axicabtagene Ciloleucel: Retreatment (MZL) (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Blindness (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 16 | 6 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Coccidioidomycosis (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 3 | 1 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 1 | 0 | 0
Mycobacterium kansasii infection (Infections and infestations) | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 10 | 3 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0
Haptoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Myeloblast count increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute bilineal leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 2 | 1 | 0 | 0
Aura (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 8 | 3 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 2 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 3 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 7 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 3 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 3 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axicabtagene Ciloleucel: Follicular Lymphoma (N=124) | Axicabtagene Ciloleucel: Marginal Zone Lymphoma (N=28) | Axicabtagene Ciloleucel: Retreatment (FL) (N=14) | Axicabtagene Ciloleucel: Retreatment (MZL) (N=2)
Anaemia (Blood and lymphatic system disorders) | 46 | 14 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 19 | 4 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 10 | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 47 | 9 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 3 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 7 | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 41 | 8 | 3 | 2
Tachycardia (Cardiac disorders) | 14 | 4 | 1 | 0
Dry eye (Eye disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 16 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 35 | 7 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 33 | 9 | 3 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 45 | 17 | 5 | 2
Vomiting (Gastrointestinal disorders) | 28 | 9 | 0 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 32 | 10 | 3 | 0
Fatigue (General disorders) | 50 | 15 | 3 | 2
Gait disturbance (General disorders) | 9 | 2 | 0 | 0
Malaise (General disorders) | 7 | 2 | 1 | 0
Oedema peripheral (General disorders) | 10 | 4 | 1 | 1
Pain (General disorders) | 17 | 3 | 0 | 1
Pyrexia (General disorders) | 99 | 24 | 8 | 2
Hypogammaglobulinaemia (Immune system disorders) | 22 | 6 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 4 | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 2 | 0 | 0
Influenza (Infections and infestations) | 3 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 9 | 4 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 10 | 4 | 0 | 0
Rhinovirus infection (Infections and infestations) | 5 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 9 | 4 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 8 | 0 | 0
Urinary tract infection (Infections and infestations) | 8 | 4 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1
Administration related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 11 | 6 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 3 | 0 | 0
Blood fibrinogen decreased (Investigations) | 3 | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 8 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 30 | 14 | 2 | 1
Platelet count decreased (Investigations) | 19 | 6 | 1 | 1
Weight decreased (Investigations) | 5 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 23 | 9 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 28 | 9 | 6 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 6 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 4 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 22 | 6 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 6 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 5 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 5 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 21 | 5 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 5 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 | 6 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 14 | 3 | 0 | 0
Disturbance in attention (Nervous system disorders) | 7 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 24 | 3 | 3 | 1
Dysgeusia (Nervous system disorders) | 3 | 3 | 0 | 0
Encephalopathy (Nervous system disorders) | 21 | 5 | 0 | 0
Headache (Nervous system disorders) | 55 | 12 | 5 | 2
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 7 | 5 | 1 | 0
Tremor (Nervous system disorders) | 35 | 8 | 2 | 1
Agitation (Psychiatric disorders) | 8 | 3 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 4 | 0 | 0
Confusional state (Psychiatric disorders) | 25 | 7 | 2 | 0
Delirium (Psychiatric disorders) | 3 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 22 | 3 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 3 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 6 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 26 | 9 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 1 | 0
Embolism (Vascular disorders) | 4 | 1 | 0 | 1
Hypertension (Vascular disorders) | 14 | 5 | 0 | 0
Hypotension (Vascular disorders) | 59 | 15 | 3 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03105336/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03105336/SAP_001.pdf